CLINICAL TRIAL: NCT04004715
Title: Effects of Protein Quality on Post-exercise Skeletal Muscle and Whole-body Protein Kinetics During Negative Energy Balance
Brief Title: Effects of Protein Quality on Post-exercise Skeletal Muscle and Whole-body Protein Kinetics During Energy Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Stefan Pasiakos, Nutritional Physiologist, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-06HC
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Whole-body Protein Balance; Muscle Protein Synthesis
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Randomized, partially-blind, cross-over controlled trial
Who Masked: Participant, Investigator
Masking Description: All participants and investigators will be blinded to the the beverage treatments. The meal treatment is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Essential Amino Acid Enriched Whey Protein (Experimental): protein powder formulation that includes whey and free-form essential amino acids
  Interventions: Dietary Supplement: Essential Amino Acid Enriched Whey Protein
- Whey Protein (Active Comparator): commercially available whey protein isolate
  Interventions: Dietary Supplement: Whey Protein
- Military Ration Entree (Active Comparator): chili and beans entree; current meal component of the meals ready to eat rations
  Interventions: Dietary Supplement: Military Ration Entree

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid Enriched Whey Protein — protein powder formulation that includes whey and free-form essential amino acids
  Arms: Essential Amino Acid Enriched Whey Protein
Dietary Supplement: Whey Protein — commercially available whey protein isolate
  Arms: Whey Protein
Dietary Supplement: Military Ration Entree — chili and beans entree; current meal component of the meals ready to eat rations
  Arms: Military Ration Entree

SUMMARY:
The optimal EAA-containing protein format necessary to maximally stimulate muscle protein synthesis and optimize whole-body net protein balance during caloric deprivation has not been determined. This study will address that gap in knowledge by examining post, whole-body exercise muscle and whole-body protein kinetic responses to ingesting varying EAA-containing protein formats after a 5 day period of negative energy balance. This study will provide the initial evidence to support the development of a recovery-based food product for military combat rations.

DETAILED DESCRIPTION:
Ten resistance-trained adults will complete this ~55-d randomized, cross-over study. Participants will participate in three, non-consecutive 5-d controlled energy deficit periods, each separated by a 14-d washout period (i.e., sufficient time to restore nitrogen and metabolic homeostasis after moderate weight loss). Post-exercise (whole-body exercise model) muscle protein synthesis (MPS) and whole-body protein turnover responses to varying EAA-containing protein formats will be determined the morning after completing the 5-d energy deficit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 35 years
* Body mass index < 30.0 kg/m2
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO) or home duty station medical support
* Resistance exercise trained defined by self-report as performing ≥ 2 sessions/wk for previous 6 mo
* Refrain from taking any nonsteroidal anti-inflammatory drugs (e.g., aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product for 10 days before starting and at least 5 days after completing the study
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes); vaping, chewing tobacco, caffeine, and dietary supplement use throughout the entire study period
* Supervisor approval for federal civilian employees and non-HRV active duty military personnel working within the US Army Natick Soldier Systems Center

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability as determined by the USARIEM or home duty station Office of Medical Support and Oversight (OMSO)
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Abnormal PT/PTT test or problems with blood clotting
* History of complications with lidocaine
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Blood donation within 8-wk of beginning the study
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test or self-report for breastfeeding will be obtained before body composition testing)
* Unwillingness or inability to consume study diets or foods provided

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
How fast participants build skeletal muscle after ingesting varying forms of essential amino acid-containing proteins after exercise | ~4.5 hour measure of muscle protein synthesis
  Assessed using stable isotope infusions of phenylalanine.

SECONDARY OUTCOMES:
How well participants suppress the degradation of body proteins while stimulating the growth of new proteins after ingesting varying forms of essential amino acid-containing proteins after exercise. | ~4.5 hour measure of whole-body protein balance
  Assessed using stable isotope infusions of tyrosine.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Pasiakos, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

REFERENCES:
- [Derived] Gwin JA, Church DD, Hatch-McChesney A, Allen JT, Wilson MA, Varanoske AN, Carrigan CT, Murphy NE, Margolis LM, Carbone JW, Wolfe RR, Ferrando AA, Pasiakos SM. Essential amino acid-enriched whey enhances post-exercise whole-body protein balance during energy deficit more than iso-nitrogenous whey or a mixed-macronutrient meal: a randomized, crossover study. J Int Soc Sports Nutr. 2021 Jan 7;18(1):4. doi: 10.1186/s12970-020-00401-5. PMID 33413462